CLINICAL TRIAL: NCT05333952
Title: A Randomized Controlled Study on the Waveform Periodicity Analysis of Complex Fractionated Electrograms in Patients With Persistent Atrial Fibrillation
Brief Title: Waveform Periodicity Analysis of Complex Fractionated Electrograms in Patients With Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-07-008C
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Catheter ablation; Mapping technique; Substrate mapping; Non-linear electrogram morphology analysis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pulmonary vein isolation + Waveform Periodicity Group (Experimental): Pulmonary vein isolation + Substrate ablation
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Substrate ablation(PRISM based)
- Pulmonary vein isolation group (Other): Pulmonary vein isolation (Conventional treatment)
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — The 3D geometry of the LA will be created using CARTO 3 system (version 6) with UDM Module and VISITAG Optimum Device Performance (ODP) module. Continuous circumferential lesions will then be created encircling the right and left PV ostia using a 7.5F, 3.5-mm Thermocool SMARTTOUCH ablation catheter (Biosense Webster, Inc., Diamond Bar, CA, USA).Pentaray catheter will be used and facilitate the high density mapping of atrial substrate (PentarayTM, Biosense Webster Inc., Diamond Bar, CA, USA). The radiofrequency energy will be applied with contact force range 5-25 g continuously with a target Ablation Index target 380-400 on the posterior wall and 550 - 600 on the anterior wall and maximum power of 25-35W in a power control mode.
Procedure: Substrate ablation(PRISM based) — Substrate modification will be guided by waveform periodicity analysis. The User Defined Map of waveform periodicity analysis will be also created by CARTO 3 system (version 6) with and VISITAG ODP module. Pentaray catheter will be used and facilitate the high density mapping of atrial substrate (PentarayTM, Biosense Webster Inc., Diamond Bar, CA, USA). Substrate modification based on waveform periodicity analysis will be performed by using a 7.5F, 3.5-mm Thermocool SMARTTOUCH ablation catheter (Biosense Webster, Inc., Diamond Bar, CA, USA). The radiofrequency energy will be applied with contact force range 5-25 g continuously with a target Ablation Index target 380-400 on the posterior wall and 550 - 600 on the anterior wall and maximum power of 25-35W in a power control mode.
  Arms: Pulmonary vein isolation + Waveform Periodicity Group

SUMMARY:
Atrial fibrillation (AF) has been the most frequently occurring, sustained arrhythmia, which causes significant morbidity and mortality. AF may not always be a totally random process. It can be maintained by stable and rapid reentrant circuits resulting in fibrillary conduction throughout the atria. During mapping of AF, difficulty is frequently encountered during the identification of culprit sites and an analysis of the wave propagation particularly when the electrogram signals demonstrate wide temporal and spatial disparities. Catheter ablation targeting regions with fractionated potentials or high frequencies during AF, has been previously proposed as a treatment strategy. However, the benefit of adjunctive CFAE (complex fractionated atrial electrogram) ablation or linear ablation after successful PVI (pulmonary vein isolation) was controversial based on the recent data from the Substrate and Trigger Ablation for Reduction of Atrial Fibrillation Trial Part II (STAR AF II) trial. Therefore, the optimal ablation strategy for persistent AF remains undetermined and an alternative approach has to be explored.

DETAILED DESCRIPTION:
In this prospective trial, investigators will investigate the long-term efficacy of catheter ablation of non-paroxysmal AF, based on selective atrial substrate modification (e.g. wavefrom periodicity analysis, similarity, plus phase mapping) (1). The control group would be PV isolation alone. The primary end point is long-term recurrence of atrial arrhythmias. The secondary end points composite procedural termination, the safety of the procedure, recurrence of multiple procedures, and change of atrial and ventricular function after catheter ablation.

The inclusion criteria, exclusion criteria, stepwise catheter ablation procedures (PVI and then substrate modification), and the follow-up procedure are the same as current treatment approaches in patients with non-paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patents who sign the informed consent forms, and allow to be followed.
2. Symptomatic AF refractory or intolerant to at least one Class 1 or 3 antiarrhythmic medication.
3. Patients with persistent/permanent AF (sustained beyond seven days, or lasting less than seven days but necessitating pharmacologic or electrical cardioversion).
4. Patients with age equal or greater than 20 years old regardless of gender.

Exclusion Criteria:

1. The presence of a atrial or ventricular thrombus.
2. Patients who are allergic to or unsuitable for use with the contrast media.
3. Pregnant patients or patients who are unavailable to receive X-ray.
4. Patients with renal insufficiency.
5. Patients had autonomic nervous system disorder (e.g. respiratory apnea) or previous catheter ablation in the LA or MAZE procedure.
6. Patients who do not need atrial substrate modification (patients with non-paroxysmal AF respond to PVI in terms of procedural termination of AF).
7. Patients with age less than 20 years old or greater than 90 years old regardless of gender.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in retention rate of normal sinus rhythm after catheter-based ablation of atrial fibrillation | Baseline and 3, 6, 9 and 12 months after catheter-based ablation of atrial fibrillation
  A 24-hour Holter monitoring and/or ECG (7 days recordings) will be performed at 3, 6, 9, and 12 months post ablation and/or when the patients experience symptoms suggestive of a tachycardia after the ablation.
  Measurements: documentation of AF signal duration more than 30 seconds.

SECONDARY OUTCOMES:
LAD | after catheter ablation of atrial fibrillation 3, 6, 12 month
  Echocardiography will be performed at 3, 6, and 12 month post-ablation for cardiac chamber dimension and atrial systolic function to assess the reverse remodeling of atrial substrate after catheter ablation of AF.
  LAD [left atrial diameter]
LVEF | after catheter ablation of atrial fibrillation 3, 6, 12 month
  Echocardiography will be performed at 3, 6, and 12 month post-ablation for cardiac chamber dimension and ventricular systolic function to assess the reverse remodeling of atrial substrate after catheter ablation of AF.
  LVEF [left ventricular ejection fraction]
e/e' | after catheter ablation of atrial fibrillation 3, 6, 12 month
  Echocardiography will be performed at 3, 6, and 12 month post-ablation for cardiac chamber dimension and ventricular systolic function to assess the reverse remodeling of atrial substrate after catheter ablation of AF.
  e/e'[the ratio of early diastolic mitral inflow velocity to early diastolic mitral annulus velocity]

CONTACTS AND LOCATIONS:
Overall Officials: Yenn-Jiang Lin, MD, PhD, Principal Investigator — Director of Cardiology Division of Taipei Veterans General Hospital
Locations (1):
- Taipei General Veterans Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The patient's data was available to the host of IRB.

REFERENCES:
- [Result] Lin CY, Lin YJ, Lo MT, Chiang CH, Chen YY, Kuo L, Chang SL, Lo LW, Hu YF, Chao TF, Chung FP, Liao JN, Chang TY, Lin C, Tuan TC, Wu CI, Liu CM, Liu SH, Cheng WH, Lugtu IC, Jain A, Ton AN, Hermanto DY, Chen SA. Efficacy of Patient-Specific Strategy: Catheter Ablation Strategy of Persistent Atrial Fibrillation Based on Morphological Repetitiveness by Periodicity and Similarity. Circ Arrhythm Electrophysiol. 2021 May;14(5):e009719. doi: 10.1161/CIRCEP.121.009719. Epub 2021 May 17. No abstract available. PMID 33998256
- [Result] Hsieh YC, Lin YJ, Lo MT, Chen YY, Lin CY, Lin C, Chung FP, Lo LW, Chang SL, Chao TF, Hu YF, Tuan TC, Liao JN, Wu CI, Liu CM, Vicera JB, Chen CC, Chin CG, Lugtu IC, Chen SA. Optimal substrate modification strategies using catheter ablation in patients with persistent atrial fibrillation: 3-year follow-up outcomes. J Cardiovasc Electrophysiol. 2021 Jun;32(6):1561-1571. doi: 10.1111/jce.15033. Epub 2021 May 5. PMID 33825268
- [Result] Lin CY, Lin YJ, Narayan SM, Baykaner T, Lo MT, Chung FP, Chen YY, Chang SL, Lo LW, Hu YF, Liao JN, Tuan TC, Chao TF, Te ALD, Kuo L, Vicera JJB, Chang TY, Salim S, Chien KL, Chen SA. Comparison of phase mapping and electrogram-based driver mapping for catheter ablation in atrial fibrillation. Pacing Clin Electrophysiol. 2019 Feb;42(2):216-223. doi: 10.1111/pace.13573. Epub 2018 Dec 27. PMID 30536679
- [Derived] Lin CY, Lin YJ, Higa S, Tsai WC, Lo MT, Chiang CH, Chang SL, Lo LW, Hu YF, Chao TF, Chung FP, Liao JN, Chang TY, Lin C, Tuan TC, Kuo L, Wu CI, Liu CM, Liu SH, Kuo MJ, Liao YC, Chuang CM, Chen YY, Hsieh YC, Chen SA. Catheter Ablation With Morphologic Repetitiveness Mapping for Persistent Atrial Fibrillation. JAMA Netw Open. 2023 Nov 1;6(11):e2344535. doi: 10.1001/jamanetworkopen.2023.44535. PMID 37991761